CLINICAL TRIAL: NCT03665207
Title: Impact of Tight Blood Glucose Control Within Normal Fasting Ranges With Insulin Titration Prescribed by the Leuven Algorithm in Adult Critically Ill Patients
Brief Title: Tight Versus Liberal Blood Glucose Control in Adult Critically Ill Patients
Acronym: TGC-fast
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other); Research Foundation Flanders (Other)
Responsible Party: Principal Investigator, Greet Van den Berghe, Full professor, Head of the clinical department and laboratory of intensive care medicine, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S61145; 2018-000756-17 (EudraCT Number)
Record Dates: First submitted 2018-08-29; First posted 2018-09-11 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Critical Illness; Hyperglycemia
MeSH Terms: conditions — Critical Illness; Hyperglycemia | interventions — Insulin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tight glucose control (Experimental): Target normal fasting blood glucose concentrations (80-110 mg/dl) with insulin therapy, administered through continuous intravenous infusion.
  Interventions: Drug: Insulin
- Liberal glucose control (Active Comparator): Tolerate hyperglycemia up to 215 mg/dl. In patients requiring insulin therapy, insulin will be titrated to target blood glucose concentrations between 180 and 215 mg/dl.
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Insulin — When blood glucose exceeds the preset target, insulin will be administered through continuous intravenous infusion. Insulin will be titrated according to frequent measurement of blood glucose and with use of the LOGIC-insulin algorithm in the experimental group. The intervention will be stopped upon ICU discharge, or until the patient is able to resume oral feeding, or until the patient no longer has a central venous catheter, whatever comes first.

SUMMARY:
Critically ill patients usually develop hyperglycemia, which is associated with an increased risk of morbidity and mortality. Controversy exists on whether targeting normal blood glucose concentrations with insulin therapy, referred to as tight blood glucose control (TGC) improves outcome of these patients, as compared to tolerating hyperglycemia. It remains unknown whether TGC, when applied with optimal tools to avoid hypoglycemia, is beneficial in a context of withholding early parenteral nutrition. The TGC-fast study hypothesizes that TGC is beneficial in adult critically ill patients not receiving early parenteral nutrition, as compared to tolerating hyperglycemia.

ELIGIBILITY:
Inclusion Criteria:

- Adult patient (18 years or older) admitted to a participating intensive care unit (ICU)

Exclusion Criteria:

* Patients with a do not resuscitate (DNR) order at the time of ICU admission
* Patients expected to die within 12 hours after ICU admission (= moribund patients)
* Patients able to receive oral feeding (not critically ill)
* Patients without arterial and without central venous line and without imminent need to place it as part of ICU management (not critically ill)
* Patients previously included in the trial (when readmission is within 48 hours post ICU discharge, the trial intervention will be resumed)
* Patients included in an IMP-RCT of which the PI indicates that co-inclusion is prohibited
* Patients transferred from a non-participating ICU with a pre-admission ICU stay >7 days
* Patients planned to receive parenteral nutrition during the first week in ICU
* Patients suffering from diabetic ketoacidotic or hyperosmolar coma on ICU admission
* Patients with inborn metabolic diseases
* Patients with insulinoma
* Patients known to be pregnant or lactating
* Informed consent refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9230 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Duration of ICU dependency | up to 1 year after randomization
  crude number of days with need for vital organ support and time to live discharge from ICU

SECONDARY OUTCOMES:
ICU Mortality | up to 1 year after randomization (with and without censoring at 90 days post randomization)
Hospital Mortality | up to 1 year after randomization (with and without censoring at 90 days post randomization)
90-day mortality | up to 90 days post randomization
Blood glucose concentrations in ICU | up to 1 year post randomization, with and without censoring at 90 days post randomization
Duration of ICU dependency | up to 90 days post randomization
  crude number of days with need for vital organ support and time to live discharge from ICU
Length of stay in hospital | up to 1 year post randomization, with and without censoring at 90 days post randomization
Time to (live) discharge from hospital | up to 1 year post randomization, with and without censoring at 90 days post randomization
Incidence of new infections in ICU | up to 1 year post randomization, with and without censoring at 90 days post randomization
Type of new infections in ICU | up to 1 year post randomization, with and without censoring at 90 days post randomization
Duration of antibiotic treatment in ICU | up to 1 year post randomization, with and without censoring at 90 days post randomization
Time course of daily C-reactive protein in ICU | up to 1 year post randomization, with and without censoring at 90 days post randomization
Time to final (live) weaning from mechanical respiratory support in ICU | up to 1 year post randomization, with and without censoring at 90 days post randomization
Number of participants with need for a tracheostomy during ICU stay | up to 1 year post randomization, with and without censoring at 90 days post randomization
Presence of clinical, electrophysiological and morphological signs of respiratory and peripheral muscle weakness in ICU | up to 1 year post randomization, with and without censoring at 90 days post randomization (in selected centers)
Incidence of acute kidney injury in ICU | up to 1 year post randomization, with and without censoring at 90 days post randomization
Duration of acute kidney injury | up to 1 year post randomization, with and without censoring at 90 days post randomization
Rate of recovery from acute kidney injury | up to 1 year post randomization, with and without censoring at 90 days post randomization
Number of participants with need for new renal replacement therapy in ICU | up to 1 year post randomization, with and without censoring at 90 days post randomization
Rate of recovery from new renal replacement therapy | up to 1 year post randomization, with and without censoring at 90 days post randomization
Number of participants with need for hemodynamic support in ICU | up to 1 year post randomization, with and without censoring at 90 days post randomization
  Hemodynamic support is defined as the need for either pharmacological (inotropes/vasopressors) and/or mechanical hemodynamic support.
Duration of hemodynamic support in ICU | up to 1 year post randomization, with and without censoring at 90 days post randomization
Time to (live) weaning from hemodynamic support | up to 1 year post randomization, with and without censoring at 90 days post randomization
Time course of markers of liver dysfunction in ICU | up to 1 year post randomization, with and without censoring at 90 days post randomization
  including transaminases, gamma-glutamyltransferase, alkaline phosphatase and bilirubin
Number of readmissions to the ICU within 48 hours after discharge | up to 1 year post randomization, with and without censoring at 90 days post randomization
Incidence of delirium in ICU (in selected centers) | up to 1 year post randomization, with and without censoring at 90 days post randomization
Rehabilitation/functional outcome | up to 2 years post randomization
  including the score obtained from the 36-item short form health survey (SF-36). The score ranges from 0 to 100, with 100 being the best possible outcome.
Rehabilitation/functional outcome in patients with brain injury | up to 1 year post randomization
  including the score obtained on the modified Rankin scale. The score ranges from 0 to 6, with 0 being the best possible outcome.
Rehabilitation/functional outcome in patients with brain injury | up to 1 year post randomization
  including the score obtained on the extended Glasgow outcome scale. The score ranges from 1 to 8, with 8 being the best possible outcome.
Blood lipid concentrations in ICU | up to 4 years post randomization (in selected centers)
Muscle strength | up to 4 years post randomization (in selected centers)
  including handgrip strength as % of the predicted value
Rehabilitation/Functional outcome | up to 4 years post randomization (in selected centers)
  including the 6-minutes walking distance in meter
Rehabilitation/Functional outcome | up to 4 years post randomization (in selected centers)
  including the score obtained from the SF-36 health survey. The score ranges from 0 to 100, with 100 being the best possible outcome.
Rate of recovery of organ function | up to 4 years post randomization (in selected centers)
Survival | up to 4 years post randomization (in selected centers)
Use of intensive care resources during index hospitalization | up to 1 year post randomization

OTHER OUTCOMES:
Biochemical markers on blood samples | up to 4 years post randomization
  including amino acid levels, blood lipid levels, cytokines, hypothalamic-pituitary hormones, glucagon, C-peptide, (epi)genetic markers
Rate of patients with muscle degeneration during ICU stay | up to 30 days post randomization (in selected centers)
  assessed by microscopy
Biochemical markers in muscle tissue during ICU stay | up to 30 days post randomization (in selected centers)
  including tissular glucose and metabolites, lipid metabolites, myofibrillary proteins, mitochondrial complex activity, autophagy markers, proteasome activity, (epi)genetic markers
Rate of patients with pathological cellular alterations in fat tissue during ICU stay | up to 30 days post randomization (in selected centers)
  assessed by microscopy
Biochemical markers in fat tissue during ICU stay | up to 30 days post randomization (in selected centers)
  including tissular glucose and metabolites, lipid metabolites, mitochondrial complex activity, autophagy markers, (epi)genetic markers
Rate of patients with muscle degeneration | up to 4 years post randomization (in selected centers)
  assessed by microscopy
Biochemical markers in muscle tissue | up to 4 years post randomization (in selected centers)
  including tissular glucose and metabolites, lipid metabolites, myofibrillary proteins, mitochondrial complex activity, autophagy markers, proteasome activity, (epi)genetic markers
Rate of patients with pathological cellular alterations in fat tissue | up to 4 years post randomization (in selected centers)
  assessed by microscopy
Biochemical markers in fat tissue | up to 4 years post randomization (in selected centers)
  including tissular glucose and metabolites, lipid metabolites, mitochondrial complex activity, autophagy markers, (epi)genetic markers

CONTACTS AND LOCATIONS:
Overall Officials: Greet Van den Berghe, MD, PhD, Study Director — KU Leuven; Jan Gunst, MD, PhD, Principal Investigator — KU Leuven
Locations (4):
- Belgium (4):
  - Department of Intensive Care Medicine, University Hospital Ghent, Ghent
  - Department of Intensive Care Medicine, Jessa Hospital Hasselt, Hasselt
  - Department of Intensive Care Medicine, University Hospitals Leuven, Leuven
  - Medical Intensive Care Unit, University Hospitals Leuven, Leuven

IPD SHARING:
Plan to Share IPD: No
Data sharing will be considered only on a collaborative basis with PIs, after evaluation of the proposed study protocol and statistical analysis plan.

REFERENCES:
- [Background] van den Berghe G, Wouters P, Weekers F, Verwaest C, Bruyninckx F, Schetz M, Vlasselaers D, Ferdinande P, Lauwers P, Bouillon R. Intensive insulin therapy in critically ill patients. N Engl J Med. 2001 Nov 8;345(19):1359-67. doi: 10.1056/NEJMoa011300. PMID 11794168
- [Background] Van den Berghe G, Wilmer A, Hermans G, Meersseman W, Wouters PJ, Milants I, Van Wijngaerden E, Bobbaers H, Bouillon R. Intensive insulin therapy in the medical ICU. N Engl J Med. 2006 Feb 2;354(5):449-61. doi: 10.1056/NEJMoa052521. PMID 16452557
- [Background] Vlasselaers D, Milants I, Desmet L, Wouters PJ, Vanhorebeek I, van den Heuvel I, Mesotten D, Casaer MP, Meyfroidt G, Ingels C, Muller J, Van Cromphaut S, Schetz M, Van den Berghe G. Intensive insulin therapy for patients in paediatric intensive care: a prospective, randomised controlled study. Lancet. 2009 Feb 14;373(9663):547-56. doi: 10.1016/S0140-6736(09)60044-1. Epub 2009 Jan 26. PMID 19176240
- [Background] NICE-SUGAR Study Investigators; Finfer S, Chittock DR, Su SY, Blair D, Foster D, Dhingra V, Bellomo R, Cook D, Dodek P, Henderson WR, Hebert PC, Heritier S, Heyland DK, McArthur C, McDonald E, Mitchell I, Myburgh JA, Norton R, Potter J, Robinson BG, Ronco JJ. Intensive versus conventional glucose control in critically ill patients. N Engl J Med. 2009 Mar 26;360(13):1283-97. doi: 10.1056/NEJMoa0810625. Epub 2009 Mar 24. PMID 19318384
- [Background] Casaer MP, Mesotten D, Hermans G, Wouters PJ, Schetz M, Meyfroidt G, Van Cromphaut S, Ingels C, Meersseman P, Muller J, Vlasselaers D, Debaveye Y, Desmet L, Dubois J, Van Assche A, Vanderheyden S, Wilmer A, Van den Berghe G. Early versus late parenteral nutrition in critically ill adults. N Engl J Med. 2011 Aug 11;365(6):506-17. doi: 10.1056/NEJMoa1102662. Epub 2011 Jun 29. PMID 21714640
- [Background] Fivez T, Kerklaan D, Mesotten D, Verbruggen S, Wouters PJ, Vanhorebeek I, Debaveye Y, Vlasselaers D, Desmet L, Casaer MP, Garcia Guerra G, Hanot J, Joffe A, Tibboel D, Joosten K, Van den Berghe G. Early versus Late Parenteral Nutrition in Critically Ill Children. N Engl J Med. 2016 Mar 24;374(12):1111-22. doi: 10.1056/NEJMoa1514762. Epub 2016 Mar 15. PMID 26975590
- [Derived] Gunst J, Debaveye Y, Guiza F, Dubois J, De Bruyn A, Dauwe D, De Troy E, Casaer MP, De Vlieger G, Haghedooren R, Jacobs B, Meyfroidt G, Ingels C, Muller J, Vlasselaers D, Desmet L, Mebis L, Wouters PJ, Stessel B, Geebelen L, Vandenbrande J, Brands M, Gruyters I, Geerts E, De Pauw I, Vermassen J, Peperstraete H, Hoste E, De Waele JJ, Herck I, Depuydt P, Wilmer A, Hermans G, Benoit DD, Van den Berghe G; TGC-Fast Collaborators. Tight Blood-Glucose Control without Early Parenteral Nutrition in the ICU. N Engl J Med. 2023 Sep 28;389(13):1180-1190. doi: 10.1056/NEJMoa2304855. PMID 37754283
- [Derived] Gunst J, Mebis L, Wouters PJ, Hermans G, Dubois J, Wilmer A, Hoste E, Benoit D, Van den Berghe G. Impact of tight blood glucose control within normal fasting ranges with insulin titration prescribed by the Leuven algorithm in adult critically ill patients: the TGC-fast randomized controlled trial. Trials. 2022 Sep 19;23(1):788. doi: 10.1186/s13063-022-06709-8. PMID 36123593